CLINICAL TRIAL: NCT05772793
Title: Usability and Adherence of Visually Impaired to Telerehabilitation: a Multicentre Study
Brief Title: Telerehabilitation for Visually Impaired
Status: Completed | Type: Observational
Sponsor: Amore Filippo (Other)
Responsible Party: Sponsor-Investigator, Amore Filippo, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 4244
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The home visual telerehabilitation path using the EyeFitness software consisted of performing one visual training session per day, 5 days a week (from Monday to Friday) for a total of 6 weeks.

SUMMARY:
the purpose of the study is to evaluate the software usability and patient's adherence from five vision rehabilitation centres. In addition, the effect and benefits of a customizable telerehabilitation program were tested.

DETAILED DESCRIPTION:
The software is used in our practice for every day vision rehabilitation training.

So it is part of our routine medical care, and a we are going to study studies the effect of the intervention in several different centers.

ELIGIBILITY:
Inclusion Criteria:

* All patients were eligible if they were over 18 years old and had a best corrected visual acuity (BCVA) between 1.3 logMAR and 0.4 LogMAR and/or a visual field of less than 60%, according to the WHO classification.

Exclusion Criteria:

* Subjects were excluded if they had a cognitive/psychiatric impairment or a motor disability that prevents the use of a computer pointing device (mouse).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients were eligible if they were over 18 years old and had a best corrected visual acuity (BCVA) between 1.3 logMAR and 0.4 LogMAR and/or a visual field of less than 60%, according to the WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Utility of EyeFitness telerehabilitation | 6 months
  The aim of this study is to evaluate the utility of the EyeFitness telerehabilitation software and the adherence of patients to the treatment.
  In order to evaluate the utility of the software the primary outcome measures were PSSUQ Version 3 scores defined as Overall, System Usefulness (Sysuse), Information Quality (Infoqual), Interface Quality (Iterqual).

SECONDARY OUTCOMES:
Effect of treatment | 6 months
  The secondary outcome measures selected for the effectiveness analysis were distance Best Corrected Visual Acuity, MNRead reading acuity, reading speed (words per minute), contrast sensitivity (at Pelli - Robson charts) and fixation stability according to Microperimeter exame classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No